CLINICAL TRIAL: NCT06501105
Title: Clinical Study to Evaluate the Performance of WOUNDCHEK Bacterial Status
Brief Title: Performance of WOUNDCHEK Bacterial Status
Status: Recruiting | Type: Observational
Sponsor: Woundchek Laboratories BV (Industry)
Collaborators: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: PROT-2023-002
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Wound Heal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- WOUNDCHEK Bacterial Status positive: Wounds positive for bacterial protease activity that may delay healing if untreated. Pre- and post-test treatment plan recorded.
  Interventions: Device: WOUNDCHEK Bacterial Status
- WOUNDCHEK Bacterial Status negative: Wounds negative for bacterial protease activity. Pre- and post-test treatment plan recorded.
  Interventions: Device: WOUNDCHEK Bacterial Status

INTERVENTIONS:
Device: WOUNDCHEK Bacterial Status — Lateral flow point of care test for the qualitative detection of bacterial protease activity in wound fluid.

SUMMARY:
The purpose of this clinical study is to evaluate the performance of WOUNDCHEK™ Bacterial Status (WCBS) when the test result is used to inform treatment decisions.

DETAILED DESCRIPTION:
The clinician treating the wound will be allowed to use the test result in treatment decisions. The pretest treatment plan will be documented on the Case Report Form (CRF) prior to performing the WCBS test. After receiving the test result the clinician will document the post-test treatment plan. The healing outcome at 12 weeks following the test will be recorded on the CRF. The study will evaluate the healing outcomes compared to when test results are not used to assist in treatment decisions with study success defined as a higher healing rate and/or mean wound size reduction for WCBS positive wounds than obtained in the study PROT-2023-001. Also, the healing rate of wounds with a negative test result will be compared to the pretest rate to ensure that clinicians do not neglect and under treat this cohort with success criteria being that the WCBS negative wound healing rate is not worse than the pre-test healing rate. Additionally, the study will establish whether there are any device related Serious Adverse Events (SAEs) or Unanticipated Adverse Device Effects (UADEs).

ELIGIBILITY:
Inclusion Criteria:

1. Subject has presented to the participating study site with a VLU, DFU and / or a PU that is suspected not to be infected, as determined by the Investigator and/ or study staff - defined as one that does not show more than two of the NERDS signs of infection.
2. Subject is 18 years of age or older.
3. The wound is between 21 days and 6 months of age or more than 6 months of age if less than 1cm2 in area.
4. Subject agrees to complete all aspects of the study and provides written Informed Consent per IRB requirements.

Exclusion Criteria:

1. Subject does not meet inclusion criteria.
2. Target wound contains a malignancy.
3. Subject has hypersensitivity of the wound or painful wound surface which prevents touching/swabbing of the wound surface.
4. Subject is confirmed to be positive for HIV or hepatitis

   .
5. Subject is unable or unwilling to provide informed consent.
6. A designated wound area may only be enrolled once in the study. For example, if an enrolled wound heals to complete closure and then re-opens, it cannot be re-enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the wound clinic with a venous leg ulcer, diabetic foot ulcer or pressure ulcer not considered to be infected and meeting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Healing rate and mean percent wound area reduction | 12 weeks
  Rate of healing and/or mean percent wound area reduction for WOUNDCHEK Bacterial Status positive wounds will be higher than obtained in the clinical study PROT-2023-001

SECONDARY OUTCOMES:
WOUNDCHEK Bacterial Status negative wound healing rate | 12 weeks
  The pre-test non-healing rate (i.e., [Non-Healed wounds/Total wounds]*100) minus the WCBS Negative wound non-healing rate (i.e. [Non-healed wounds with a negative WCBS result/Total wounds]*100) will be less than or equal to zero.
Adverse events | 12 weeks
  There will be no device related serious adverse events (SAE) or unanticipated adverse device effects (UADE).

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health Comprehensive Wound Healing & Hyperbaric Center, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.